CLINICAL TRIAL: NCT07188077
Title: Differential Analysis of Primary Central Nervous System Diffuse Large B-Cell Lymphoma Based on Metabolomics and Immunomics
Brief Title: Metabolic and Immunomic Differential Analysis of Primary Central Nervous System Diffuse Large B-Cell Lymphoma
Status: Recruiting | Type: Observational
Sponsor: Ting YANG (Other)
Responsible Party: Sponsor-Investigator, Ting YANG, Administrative Director of the Department, Fujian Medical University
Organization: Fujian Medical University (Other)
Other Study IDs: PCNSL-IMMS-01
Record Dates: First submitted 2025-09-08; First posted 2025-09-23 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Primary Central Nervous System Lymphoma (PCNSL); Diffuse Large B-Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- PCNSL: Primary Diffuse Large B-Cell Lymphoma of the Central Nervous System
- GDLBCL: Diffuse large B-cell lymphoma of the gastrointestinal tract
- DLBCL: Non-Hodgkin's diffuse large B-cell lymphoma not involving the central nervous system or gastrointestinal tract
- Health: Healthy control

SUMMARY:
This study is a prospective cohort study. The case group will include patients with primary central nervous system lymphoma confirmed by imaging and pathology. The control group will include patients with pathologically confirmed diffuse large B-cell lymphoma who have been excluded from central nervous system involvement, as well as age- and gender-matched healthy volunteers (hematopoietic stem cell donors). Baseline data (as described below) will be collected. Patients with primary CNS lymphoma will undergo follow-up every 3 months, with immediate follow-up if clinical symptoms arise.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 18 and 75 years.
2. The case group must have a confirmed diagnosis of primary central nervous system lymphoma (PCNSL) and must not have received any antitumor therapy prior to baseline sample collection.
3. Must sign an informed consent form, agree to participate in this study, and provide samples and clinical information as required.
4. Case group patients must have complete supporting imaging and pathology data.

Exclusion Criteria:

1. Presence of other systemic malignancies.
2. Presence of severe infections or metabolic disorders.
3. Use of antimetabolites or chemotherapy drugs within one week prior to sample collection.
4. Pregnant or lactating women.
5. Concurrent severe internal medical conditions (e.g., end-stage renal disease, heart failure, liver failure).
6. Patients unable to complete study requirements due to psychiatric disorders or cognitive impairment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Hematopoietic stem cell donor
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Metabolomics | Before the start of the first treatment cycle, at the end of each treatment cycle(each cycle is 28 days)
  Detection of metabolites in plasma using liquid chromatography-mass spectrometry (LC-MS) technology
CYTOF | Before the start of the first treatment cycle, at the end of each treatment cycle(each cycle is 28 days)
  Immunophenotyping of PBMCs using flow cytometry mass spectrometry (CYTOF)

SECONDARY OUTCOMES:
OS | From date of randomization until the date of the end of follow-up or date of death from any cause, whichever came first, assessed up to 12months
  Overall survival
PFS | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 12months
  Progression-free survival

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: Undecided
Protect patient privacy